CLINICAL TRIAL: NCT02033031
Title: Treatment With Anti-vascular Endothelial Growth Factor in Patients With Branch Retinal Vein Occlusion: 5 Years of Clinical Experience
Brief Title: Long-term Treatment Effect of Intravitreal Ant-VEGF in Branch Retinal Vein Occlusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Prof. Dr, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Sacu
Record Dates: First submitted 2014-01-02; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Branch Retinal Vein Occlusion
Keywords: branch retinal vein occlusion; central retinal thickness; visual acuity; central reintal sensitivity
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lucentis (Active Comparator): PRN intravitreal injection of Lucentis
  Interventions: Drug: Lucentis intravitreal injection
- Avastin (Active Comparator): PRN intravitreal injection of Lucentis
  Interventions: Drug: Avastin intravitreal injection

INTERVENTIONS:
Drug: Lucentis intravitreal injection — Lucentis intravitreal injection
  Arms: Lucentis
Drug: Avastin intravitreal injection — Avastin intravitreal injection
  Arms: Avastin

SUMMARY:
Retinal vein occlusion (RVO) is the second leading cause of retinal vascular disease in patients older than 50 years.The prevalence varies from 0.7% to 1.6% in the literature.

Visual recovery depends on ischemic damage of the retina, the occurence of macular edema (ME) and the development of neovascular glaucoma. The occurence of ME is the main reason for visual loss and frustrates visual recovery among patients with both central or branch RVO.

Therapeutic options that have been used and discussed over the years are the treatment with anticoagulants, fibrinolytics, corticosteroids, acetazolamide and isovolemic haemodilution. Furthermore, surgical options like vitrectomy and radial optic neurotomy were used. Panretinal photocoagulation and grid pattern photocoagulation had established as additional tool to induce chorioretinal anastomosis. Nevertheless, the effectiveness and the evidence of these different treatment options could not be verified and remains mostly unknown.

Nowadays, intravitreal anti-VEGF application had become the treatment of choice for ME secondary to RVO. Multi-center studies have already shown the effectiveness of anti-VEGF treatment to reduce intraretinal fluid and retinal hemorrhages (BRAVO, CRUISE). Unfortunately, often high numbers of re-treatments become necessary over the years. In our knowledge, there are no reports showing more than 3 years treatment effects of antiangiogenic drugs in patients with BRVO. However, the results of treatment effect longer than 3 years are important, as the mean age < 70 years with an onset of BRVO has been estimated in about 60% of all cases. In addition, most patients with regard to the application of anti-VEGF treatment in real clinical setting, there is only rare experience concerning need of optimum time duration for follow-up at the departments. Hence, the present study aimed to evaluate the long-term clinical outcomes, safety and therapeutic benefit of a flexible dosing regimen of intravitreal anti-VEGF therapy in patients with ME secondary to BRVO.

DETAILED DESCRIPTION:
This cross-sectional study evaluates a series of patients with ME due to RVO who were available for at least 4 years' follow-up examination. The patients received either intravitreal ranibizumab (IVR) or bevacizumab (IVB) in a flexible dosing regimen

ELIGIBILITY:
Inclusion Criteria:

* Macular edema secondary to Branch retinal vein occlusion

Exclusion Criteria:

* Aphakia, Glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
visual acuity | up to 6 months
  measurement of visual acuity outcomes; baseline in comparison to long-term

SECONDARY OUTCOMES:
retinal sensitivity | up to 6 months
  course of retinal sensitivity within the groups
central retinal thickness | up to 6 months
  course of central retinal thickness
treatment rate | up to 6 months
  treatment rate within the groups

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sacu, Prof., Principal Investigator — Medical University of Vienna, Department of Ophthalmology and Optometry
Locations (1):
- Medical University of Vienna, Vienna, Austria